CLINICAL TRIAL: NCT02987816
Title: Learning Enhancement Using Transcranial Stimulation, Leading Expertise, Acquisition and Retention of Neurosurgical Skills
Brief Title: Neurosurgical Skill Enhancement Using Transcranial Stimulation
Acronym: LETS-LEARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Patrick Ciechanski, PhD Candidate (Neurosciences), University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REB 15-2443
Record Dates: First submitted 2016-11-25; First posted 2016-12-09 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Neurosurgery
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham tDCS (Sham Comparator): Sham tDCS. 45 second ramp up to 1milliamp, 60 second current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned over the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Interventions: Device: Sham tDCS
- Anodal tDCS (Experimental): Anodal tDCS. 45 second ramp up to 1milliamp, 20 minute current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned over the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Interventions: Device: Anodal tDCS

INTERVENTIONS:
Device: Sham tDCS — NeuroConn Direct-Current Stimulator. Sham tDCS: 45 second ramp up to 1milliamp, 60 second current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned over the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Other Names: Sham transcranial direct current stimulation
  Arms: Sham tDCS
Device: Anodal tDCS — NeuroConn Direct-Current Stimulator. Sham tDCS: 45 second ramp up to 1milliamp, 20 minute current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned over the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Other Names: Anodal transcranial direct current stimulation
  Arms: Anodal tDCS

SUMMARY:
Recent changes in medical training environments and restrictive work-hour regulations have greatly impacted trainees, limiting the number of opportunities to gain proficiency in procedural skills. Reports suggest that medical residents lack confidence in their ability to perform certain medical procedures, and program directors often do not believe their residents can operate independently in major procedures. Simulator based task training (SBTT) has provided a safe and ethically appropriate method of skill acquisition but training opportunities remain limited. Methods to enhance motor learning during these training opportunities have not been described. Transcranial direct-current stimulation (tDCS) is an emerging form of non-invasive brain stimulation that has been shown to improve motor learning. tDCS has been shown to enhance increasingly complex skill acquisition. The investigators propose to examine if tDCS can improve the acquisition and retention of neurosurgical skill. The investigators propose a double blind, sham-controlled randomized trial applying tDCS during evidence-based SBTT of medical students, to determine if brain stimulation can enhance training skill acquisition and retention. Even a modest enhancement carries the potential to transform medicosurgical skills training.

DETAILED DESCRIPTION:
Rationale: Recent changes in medical training environments have resulted in many trainees lacking sufficient opportunity to acquire specific skills necessary for their specialty. New methods to enhance the acquisition and retention of medical and surgical skills are required to ensure the quality of the future physician workforce. Transcranial direct-current stimulation (tDCS) is an emerging method of non-invasive brain stimulation that has been show to safely enhance motor learning in adults and children. Even a modest enhancement of acquisition and retention of medical-surgical skill with tDCS carries the potential to accelerate skill training for health care providers, thereby contributing to greater training efficiency and improved patient outcomes.

Objectives: The objective of this study is to assess whether tDCS can enhance the acquisition and retention of neurosurgical ability.

Ethics:This study has been approval by the University of Calgary Research Ethics Board

Design: Randomized, double blind, sham-controlled trial to evaluate the ability of tDCS to enhance learning and retention of neurosurgical skills.

Transcranial Direct-Current Stimulation: The tDCS methods used are based on best-available evidence and practices, and will be applied in a standardized fashion by experienced investigators. Anodal tDCS will be delivered through saline-soaked sponge electrodes using a NeuroConn Direct-Current Stimulator (NeuroConn, Ilmenau, Germany). The anode will be centered over the left primary motor cortex (localized using the 10-20 EEG System), with the cathode over the contralateral supraorbital area. Both anodal and sham tDCS groups will have the current ramped-up to 1milliamp over 30 seconds. In the anodal tDCS group, the current will be held for 20 minutes. In the sham tDCS condition, the current will be held for only 60 seconds (no changes in cortical excitability) followed by a 30 second ramp-down.

Participants: Medical students (years 1-3) from the Cumming School of Medicine (University of Calgary) will be recruited. To ensure comparable baseline skills, trainees will be excluded if they have undergone formal neurosurgical training in the past 3 months.

Sample size calculations are based on the performance measures for the percentage of virtual tumor resected, determined through pilot studies. Based on 20% more tumor being resected at post-training, power of 90% and type-1 error of 0.05, the investigators estimate a sample size of a minimum of 24 participants (n=12 per stimulation condition).

Study Design: A short questionnaire will be completed to determine demographic characteristics, including: gender, age, level of training, how many times participants have performed on a virtual surgical simulator, how often participants play video games, and how often participants play a musical instrument.

Participants will be recruited at the Project NeuroArm Laboratory (University of Calgary) and be oriented to the workspace. Participants will complete virtual tumor resections on a NeuroTouch (National Research Council of Canada) surgical simulator. Participants will view a standardized training video, created by an expert in neurosurgery, demonstrating a virtual tumor resection using the simulator. Participant will have 3 minutes to resect a virtual tumor, avoiding resection of healthy tissue. Recorded outcome metrics will include: % tumor resected, volume of healthy tissue resected, time of excessive force on tumor and time of excessive force on healthy tissue.

Participants will perform one resection at baseline, establishing baseline skill. Participants will be randomized to receive sham or active tDCS by blinding selecting a code from the envelope, corresponding to a particular stimulation condition. Participants will perform eight training repetitions, taking approximately 30 minutes. Following approximately 30 minutes of training (eight training repetitions) the tDCS electrodes will be removed, and a final resection will be performed. Six weeks following the training the participants will return to assess retention of skill, performing a single resection. Emerging evidence suggests that a significant decay in surgical skill is present six weeks following training.

Data Analysis: Independent samples t-test will evaluate difference in outcome metrics at post-training between stimulation conditions. Two-way repeated-measures ANOVA for factors "stimulation type" and "training block" will explore the interaction between tDCS and training for each outcome metric. Retention of skill will be assessed using a paired t-test for each stimulation group.

ELIGIBILITY:
Inclusion Criteria:

* Medical student
* Informed consent

Exclusion Criteria:

* Diagnosis of a developmental, neurological or neuropsychiatric disorder
* Taking neuropsychotropic medication
* Has an irremovable implanted metal object in the head
* Has a pacemaker or other implanted electrical device
* Pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in % tumor resected | Baseline and immediately post-training
  A "baseline" trial will be performed, followed by 8 consecutive "training" trials (approximately 30 minutes of training), immediately followed by a "post-training" trial.

SECONDARY OUTCOMES:
Change in volume of healthy tissue resected | Baseline and immediately post-training
  A "baseline" trial will be performed, followed by 8 consecutive "training" trials (approximately 30 minutes of training), immediately followed by a "post-training" trial.
Change in time of excessive forces on tumor | Baseline and immediately post-training
  A "baseline" trial will be performed, followed by 8 consecutive "training" trials (approximately 30 minutes of training), immediately followed by a "post-training" trial.
Change in time of excessive forces on healthy tissue | Baseline and immediately post-training
  A "baseline" trial will be performed, followed by 8 consecutive "training" trials (approximately 30 minutes of training), immediately followed by a "post-training" trial.

OTHER OUTCOMES:
Retention of primary and secondary outcomes measures | 6 weeks following training
  Retention of skill will be examined 6 weeks following the training session. A single repetition of the tumor resection task will be performed. % tumor resected, volume of healthy tissue resected, time of excessive forces on tumor, and time of excessive forces on healthy tissue will be recorded and compared to the "post-training" trial (immediately following training).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coleman JJ, Esposito TJ, Rozycki GS, Feliciano DV. Early subspecialization and perceived competence in surgical training: are residents ready? J Am Coll Surg. 2013 Apr;216(4):764-71; discussion 771-3. doi: 10.1016/j.jamcollsurg.2012.12.045. PMID 23521960
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Reis J, Fritsch B. Modulation of motor performance and motor learning by transcranial direct current stimulation. Curr Opin Neurol. 2011 Dec;24(6):590-6. doi: 10.1097/WCO.0b013e32834c3db0. PMID 21968548
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589